CLINICAL TRIAL: NCT04035733
Title: A Phase IIa Open-label Single Arm Study of Safety and Efficacy of rVA576 in Adult Mild to Moderate Bullous Pemphigoid Subjects
Brief Title: rVA576 in Adult Mild to Moderate Bullous Pemphigoid Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AKARI Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK801
Record Dates: First submitted 2019-04-12; First posted 2019-07-29 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2021-06

CONDITIONS: Bullous Pemphigoid (BP)
MeSH Terms: conditions — Pemphigoid, Bullous

STUDY DESIGN:
Intervention Model Description: A Phase IIa open-label single arm study of safety and efficacy of rVA576 in adult mild to moderate Bullous Pemphigoid subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open-label single arm study (Experimental)
  Interventions: Drug: rVA576

INTERVENTIONS:
Drug: rVA576 — BP subjects will be treated with 30 mg once daily rVA576 regime for 6 weeks.

SUMMARY:
Bullous pemphigoid (BP) is the most common of the autoimmune blistering skin diseases in Western Europe. [Joly 2012]The study will recruit the new onset or relapsing mild to moderate BP patients. The study population will consist of patients above the age of 18 years with an active episode of BP, confirmed by inclusion and exclusion criteria and who, in the opinion of the Investigator, would benefit from treatment with rVA576. Recombinant rVA576 is a small protein complement C5 and LTB4 inhibitor, which prevents the cleavage of C5 by C5 convertase and thereby inhibits generation of C5b-9 the membrane attack complex (MAC), as well as preventing the release of the anaphylatoxin C5a. rVA576 is effective in inhibiting terminal complement activity irrespective of the activating pathway (classical, lectin or alternative). This Phase IIa open-label single-arm study will evaluate the safety and efficacy of rVA576 in adult mild to moderate Bullous Pemphigoid patients

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female ≥18-year-old patients
2. Subject with newly presenting mild to moderate cutaneous bullous pemphigoid (BP)
3. BPDAI global score at the screening of 10-56 (≥ 10 but <56)
4. Subjects with a relapse of mild to moderate bullous pemphigoid are eligible if their disease was quiescent for at least 2 months before the current relapse.
5. Cutaneous bullous pemphigoid (BP) per standard diagnostic criteria:

   1. Clinical presentation (cutaneous blistering and/or itchy dermatosis), AND
   2. Direct immunofluorescence (DIF) studies.
6. Karnofsky performance status ≥ 60%
7. Adequate cardiac, renal, hepatic, neurological and psychiatric function as determined by the Investigator and demonstrated by screening laboratory evaluations, vital sign measurement, ECG recording and physical examination results.
8. Women of childbearing potential (WOCBP) must agree to use effective contraception consistently throughout the study and have a negative serum pregnancy test at screening and a negative urine pregnancy test per the schedule of visits.
9. Males with a childbearing potential partner must agree to use effective contraception consistently OR have had a vasectomy
10. Willing and able to adhere to the study visit schedule and other protocol requirements.
11. Willing and able to provide voluntary written informed consent
12. Willing to receive immunisation against Neisseria meningitidis and antibiotic prophylaxis in accordance with applicable guidelines and local standard of care of the PI at the trial site

Exclusion Criteria:

1. Patients with severe BP. Severe disease to defined as global BPDAI ≥ 56.
2. Patients with refractory BP.
3. Suspected drug-induced BP
4. Concomitant skin conditions preventing physical evaluation of BP.
5. Participation in a clinical trial of an investigational product within 6 weeks of screening.
6. Known hypersensitivity to tick or to rVA576 and any of its excipients.
7. BP patients on systemic corticosteroid or systemic immunomodulator or other treatment for the current BP episode (including azathioprine, dapsone, doxycycline, etc) provided the treatment cannot be discontinued before Day 1.
8. Treatment with biologics (e.g. etanercept, adalimumab, ustekinumab, infliximab, intravenous immunoglobulin (IVIG) and rituximab or other anti-CD20 therapies) within 5 half-lives of the drugs prior to screening.
9. Known hypersensitivity to mometasone furoate or to other corticosteroids or to any excipients in mometasone furoate
10. Received rVA576 for the treatment of the current episode of BP prior to study entry.
11. Patients with severe medical or surgical conditions at screening or Day 1 including, but not limited to cardiac, respiratory, renal, hepatic, haematological, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, cerebral, psychiatric, or any other severe acute or chronic medical condition that may increase the risk associated with study participation/treatment or may interfere with the interpretation of study results and, in the Investigator's opinion, would make the patient inappropriate for study entry.
12. Presence of any malignancy that has been under active treatment or in previous 5 years except for patients with the removal of uncomplicated basal cell carcinoma or cutaneous squamous cell carcinoma, who may take part in the study.
13. Congenital or acquired immunodeficiency (e.g. common variable immunodeficiency, organ transplantation).
14. Clinically significant vital sign measurements or ECG findings as determined by the Investigator.
15. Clinically significant abnormal laboratory test results.
16. The active or recent history of clinically significant infection within 1 month of Screening.
17. Pregnant or breast-feeding, or planning to become pregnant during the study.
18. Evidence of an active disease of hepatitis B (HBsAg positive or HBcAg positive) or hepatitis C (HCV ab positive), CMV (IgM positive) or human immunodeficiency virus (HIV) infection (HIV1/2 Ab positive)
19. Active abuse of alcohol or drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-04-29 (Actual)

PRIMARY OUTCOMES:
Safety parameter | 42 days
  Proportion of participants reporting grade 3, 4 and 5 adverse events, which are related/possibly related to rVA576 during the treatment period.
  Treatment emergent adverse events (TEAEs) consist of:
  * Change from baseline in physical examination
  * ECG
  * Clinical laboratory tests
  * Vital signs The Common Terminology Criteria for Adverse Events (CTCAE v4.03) will be used to grade adverse events.

SECONDARY OUTCOMES:
Efficacy Parameter | 42 days
  Change in BPDAI between baseline (Day 1) and Day 42.
Quality of life questionnaire | 42 days
  Change in quality of life questionnaire between baseline (Day 1) and Day 42

CONTACTS AND LOCATIONS:
Locations (2):
- University of Lubeck, Lübeck, Germany
- UMCG Groningen, Groningen, Hanzeplein 1, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sadik CD, Rashid H, Hammers CM, Diercks GFH, Weidinger A, Beissert S, Schauer F, Fettiplace J, Thaci D, Ngai Y, Nunn MA, Zillikens D, Horvath B. Evaluation of Nomacopan for Treatment of Bullous Pemphigoid: A Phase 2a Nonrandomized Controlled Trial. JAMA Dermatol. 2022 Jun 1;158(6):641-649. doi: 10.1001/jamadermatol.2022.1156. PMID 35507334